CLINICAL TRIAL: NCT05513352
Title: Exploiting the Potential of Neural Attentional Control to Overcome Hearing Impairment
Acronym: NeurAttContr
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University of Luebeck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AuditoryAttention; 201864 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2022-08-17; First posted 2022-08-24 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Hearing Loss; Attention Impaired; Tinnitus
Keywords: neuromodulation; auditory attention; neurobiology of language; electroencephalography; transcranial alternating current stimulation; neurofeedback; alpha oscillations; speech tracking
MeSH Terms: conditions — Hearing Loss; Tinnitus

STUDY DESIGN:
Intervention Model Description: Experiment 1:
  * between-subject design
  * 3x4 = 3(hearing group) x 4(condition)
  * Masking: Single (Participant)
  * Masking Description: single-blind
  Experiment 2:
  * between-subject design
  * 3x4 = 3(hearing group) x 4(condition)
  * Masking: Single (Participant)
  * Masking Description: single-blind
  Experiment 3:
  * between-subject design
  * 3x2x2x4 = 3(hearing group) x 2 (stimulation) x 2(timepoint) x 4(condition)
  * Masking: Double (Participant, investigator)
  * Masking Description: double-blind
  Experiment 4:
  * between-subject design
  * 3x2x2x4 = 3(hearing group) x 2 (stimulation) x 2(timepoint) x 4(condition)
  * Masking: Double (Participant, investigator)
  * Masking Description: double-blind
  Experiment 5:
  * within-subject design
  * 2x2x4 = 2 (training) x 2(timepoint) x 4(condition)
  * Masking: Double (Participant, investigator)
  * Masking Description: double-blind
  Primary Purpose: Basic Science
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: single-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (19):
- Experiment 1 - Normal hearing - AAT (No Intervention): Each participant assigned to the normal hearing group will undergo one experimental session during which EEG is recorded while participants perform an auditory attention task (AAT).
- Experiment 1 - Hearing impaired - AAT (No Intervention): Each participant assigned to the normal hearing impaired group will undergo one experimental session during which EEG is recorded while participants perform an auditory attention task (AAT).
- Experiment 2 - normal hearing _ SAT (No Intervention): Each participant assigned to the normal hearing group will undergo one experimental session in which EEG is used to measure neural speech tracking while participants undergo the selective speech attention task (SAT).
- Experiment 2 - hearing impaired - SAT (No Intervention): Each participant assigned to the hearing impaired group will undergo one experimental session in which EEG is used to measure neural speech tracking while participants undergo the selective speech attention task (SAT).
- Experiment 2 - tinnitus - SAT (No Intervention): Each participant assigned to the tinnitus group will undergo one experimental session in which EEG is used to measure neural speech tracking while participants undergo the selective speech attention task (SAT).
- Experiment 3 - normal hearing (tACS) - AAT (Experimental): The subjects assigned to the normal hearing group will undertake 20min tACS stimulation applied over the temporo-parietal cortex.
  Each session will include the following three phases: (1) pre-stimulation baseline, (2) brain stimulation, and (3) post-stimulation. AAT will be conducted in each phase and concurrent EEG will be recorded.
  Interventions: Device: tACS - transcranial alternating current stimulation
- Experiment 3 - normal hearing (sham) - AAT (Sham Comparator): The subjects assigned to the normal hearing group will undertake 20min sham stimulation applied over the temporo-parietal cortex.
  Each session will include the following three phases: (1) pre-stimulation baseline, (2) sham brain stimulation, and (3) post-stimulation. AAT will be conducted in each phase and concurrent EEG will be recorded.
  Interventions: Device: sham - transcranial alternating current stimulation
- Experiment 3 - hearing impaired (tACS) - AAT (Experimental): The subjects assigned to the hearing impaired group will undertake 20min tACS stimulation applied over the temporo-parietal cortex.
  Each session will include the following three phases: (1) pre-stimulation baseline, (2) brain stimulation, and (3) post-stimulation. AAT will be conducted in each phase and concurrent EEG will be recorded.
  Interventions: Device: tACS - transcranial alternating current stimulation
- Experiment 3 - hearing impaired (sham) - AAT (Sham Comparator): The subjects assigned to the hearing impaired group will undertake 20min sham stimulation applied over the temporo-parietal cortex.
  Each session will include the following three phases: (1) pre-stimulation baseline, (2) sham brain stimulation, and (3) post-stimulation. AAT will be conducted in each phase and concurrent EEG will be recorded.
  Interventions: Device: sham - transcranial alternating current stimulation
- Experiment 3 - tinnitus (tACS) - AAT (Experimental): The subjects assigned to the tinnitus group will undertake 20min tACS stimulation applied over the temporo-parietal cortex.
  Each session will include the following three phases: (1) pre-stimulation baseline, (2) brain stimulation, and (3) post-stimulation. AAT will be conducted in each phase and concurrent EEG will be recorded.
  Interventions: Device: tACS - transcranial alternating current stimulation
- Experiment 3 - tinnitus (sham) - AAT (Sham Comparator): The subjects assigned to the tinnitus group will undertake 20min sham stimulation applied over the temporo-parietal cortex.
  Each session will include the following three phases: (1) pre-stimulation baseline, (2) sham brain stimulation, and (3) post-stimulation. AAT will be conducted in each phase and concurrent EEG will be recorded.
  Interventions: Device: sham - transcranial alternating current stimulation
- Experiment 4 - normal hearing (tACS) - SAT (Experimental): The subjects assigned to the normal hearing group will undertake 20min tACS stimulation applied over the temporo-parietal cortex.
  Each session will include the following three phases: (1) pre-stimulation baseline, (2) brain stimulation, and (3) post-stimulation. SAT will be conducted in each phase and concurrent EEG will be recorded.
  Interventions: Device: tACS - transcranial alternating current stimulation
- Experiment 4 - normal hearing (sham) - SAT (Sham Comparator): The subjects assigned to the normal hearing group will undertake 20min sham stimulation applied over the temporo-parietal cortex.
  Each session will include the following three phases: (1) pre-stimulation baseline, (2) sham brain stimulation, and (3) post-stimulation. SAT will be conducted in each phase and concurrent EEG will be recorded.
  Interventions: Device: sham - transcranial alternating current stimulation
- Experiment 4 - hearing impaired (tACS) - SAT (Experimental): The subjects assigned to the hearing impaired group will undertake 20min tACS stimulation applied over the temporo-parietal cortex.
  Each session will include the following three phases: (1) pre-stimulation baseline, (2) brain stimulation, and (3) post-stimulation. SAT will be conducted in each phase and concurrent EEG will be recorded.
  Interventions: Device: tACS - transcranial alternating current stimulation
- Experiment 4 - hearing impaired (sham) - SAT (Sham Comparator): The subjects assigned to the hearing impaired group will undertake 20min sham stimulation applied over the temporo-parietal cortex.
  Each session will include the following three phases: (1) pre-stimulation baseline, (2) sham brain stimulation, and (3) post-stimulation. SAT will be conducted in each phase and concurrent EEG will be recorded.
  Interventions: Device: sham - transcranial alternating current stimulation
- Experiment 4 - tinnitus (tACS) - SAT (Experimental): The subjects assigned to the tinnitus group will undertake 20min tACS stimulation applied over the temporo-parietal cortex.
  Each session will include the following three phases: (1) pre-stimulation baseline, (2) brain stimulation, and (3) post-stimulation. SAT will be conducted in each phase and concurrent EEG will be recorded.
  Interventions: Device: tACS - transcranial alternating current stimulation
- Experiment 4 - tinnitus (sham) - SAT (Sham Comparator): The subjects assigned to the tinnitus group will undertake 20min sham stimulation applied over the temporo-parietal cortex.
  Each session will include the following three phases: (1) pre-stimulation baseline, (2) sham brain stimulation, and (3) post-stimulation. SAT will be conducted in each phase and concurrent EEG will be recorded.
  Interventions: Device: sham - transcranial alternating current stimulation
- Experiment 5 - normal hearing (NF right) - AAT (Experimental): Each participant of the normal hearing group will undergo the neurofeedback training in which the participants learn to increase alpha power in the right relative to the left parietal cortex. Before and after the NF training, participants will perform the AAT and concurrent EEG will be recorded.
  Interventions: Device: NF - Neurofeedback
- Experiment 5 - normal hearing (NF left) - AAT (Active Comparator): Each participant of the normal hearing group will undergo the neurofeedback training in which the participants learn to increase alpha power in the left relative to the right parietal cortex. Before and after the NF training, participants will perform the AAT and concurrent EEG will be recorded.
  Interventions: Device: NF - Neurofeedback

INTERVENTIONS:
Device: tACS - transcranial alternating current stimulation — TACS is a non-invasive brain stimulation (NIBS) techniques that belong to the class of low current transcranial electric stimulation. In contrast to the better known transcranial direct current stimulation (tDCS), the tACS current is not constant, but alternates with a certain frequency.
  The stimulation will be applied over the left temporo-parietal cortex at participants' individual alpha frequency. The stimulation intensity will be 2 milliampere (mA, peak-to-peak value, corresponding to a sine wave of ±1 mA amplitude). Stimulation will be delivered through conductive rubber electrodes.
  Arms: Experiment 3 - hearing impaired (tACS) - AAT; Experiment 3 - normal hearing (tACS) - AAT; Experiment 3 - tinnitus (tACS) - AAT; Experiment 4 - hearing impaired (tACS) - SAT; Experiment 4 - normal hearing (tACS) - SAT; Experiment 4 - tinnitus (tACS) - SAT
Device: sham - transcranial alternating current stimulation — During "sham stimulation" (placebo), tACS will be ramped up and down for 12 seconds , that is, no electric stimulation wil be applied during the actual experiment. The up and down ramping will be repeated at the end of the experiment.
  The sham condition serves to evoke sensations associated with tACS stimulation, but without stimulating during the actual experiment.
  Arms: Experiment 3 - hearing impaired (sham) - AAT; Experiment 3 - normal hearing (sham) - AAT; Experiment 3 - tinnitus (sham) - AAT; Experiment 4 - hearing impaired (sham) - SAT; Experiment 4 - normal hearing (sham) - SAT; Experiment 4 - tinnitus (sham) - SAT
Device: NF - Neurofeedback — Neurofeedback (NF) is a non-invasive approach that combines neurophysiological recordings with real-time sensory feedback (most studies use visual feedback). Through real-time NF, individuals thus can learn to regulate their brain activity.
  In this study, NF will be based on concurrent EEG recordings. During NF, participants will observe a space ship automatically navigating through a narrow tunnel. The modulation of their neural alpha power lateralization into the trained direction will be rewarded by the acceleration of the space ship, a modulation in the opposite direction will reduce speed and autopilot accuracy.
  Arms: Experiment 5 - normal hearing (NF left) - AAT; Experiment 5 - normal hearing (NF right) - AAT

SUMMARY:
This study will improve the understanding of the cerebral mechanisms that underlie the control of auditory selective attention and evaluate the potential of neuromodulation to enhance neural attention control as a possible way to overcome hearing impairment.

First, electroencephalography (EEG) will be applied to identify neural marker of auditory attention in individuals with hearing loss (HL), tinnitus (TI) and normal hearing (NH). Afterwards, the importance of the identified markers for attention control will be tested using non-invasive transcranial alternating current stimulation (tACS) and neurofeedback (NF).

DETAILED DESCRIPTION:
Hearing loss and associated conditions such as tinnitus are the fourth highest cause of disability worldwide, with estimated annual cost of over 750 billion dollars. Due to the rise and ageing of the global population, the number of people with hearing impairment is growing at a rapid pace. Besides, the incidence of noise induced hearing impairment is also increasing in younger populations. A common complaint of hearing impaired individuals is the significant decline of speech comprehension under challenging listening conditions. These situations typically include reverberations, background noise or multiple speakers and they require the listener to direct attention selectively to a target sound source (e.g. the interlocutor) and to suppress distracting sounds in the background (e.g. from not attended speakers).

Auditory prostheses with pinna-imitating microphones can improve the localization of a target sound source through the sensory enhancement of spatial cues in the acoustic signal. However, the benefit of additional sensory information is limited due of the missing implementation of attention control that would permit the selective amplification of the target sound source and the suppression of irrelevant distracting noise.

The question of how the brain instantiates attentional filter mechanisms that control target amplification and distractor suppression has drawn a lot of interest in the field of cognitive neuroscience. Neural markers of auditory attention such as lateralized oscillatory brain activity in the alpha frequency band (~8-12Hz) and the enhanced neural tracking of attended of attended speech have been linked to the top-down control of attention. However, the interrelationship between these neural markers is still underexplored. Further, the functional role of alpha band oscillations in auditory attention is underspecified as they could potentially implement target enhancement and distractor suppression. Together, this limits the understanding of the neuro-cognitive basis of attention.

The proposed project aims to address this problem by improving the investigators understanding of the cerebral mechanisms that underlie the control of auditory selective attention. The outlined research project will test the hypothesis that individuals with hearing impairment have deficits in auditory distractor inhibition that are reflected by ineffective neural suppression of irrelevant information. This hypothesis will be examined in three different lines of research. In research line 1, I will test a new framework in individuals who suffer from sensorineural hearing loss or tinnitus that allows to dissociate target selection and distractor suppression at the neural level based on electroencephalography (EEG) recordings. In research lines 2-3, I will then evaluate the potential of electric brain stimulation and neurofeedback to enhance auditory distractor suppression.The results of this project will have theoretical implications for current models of auditory attention and speech comprehension by specifying the functional role of oscillatory brain activity in normal hearing individual and hearing impaired populations. Beyond, this research will contribute new insights how the control of auditory selective attention could be implemented in a brain-computer interface.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 / 55-75
* German as first language
* Normal or corrected to normal vision
* Right-handed
* Normal hearing, hearing impairment or tinnitus (see specified inclusion)
* Normal hearing: ≤20 decibel (dB) hearing level (HL) at frequencies from 250 Hz to 8,000 Hz for both ears.

Specified inclusion for Experiment 1, 2, 3 & 4:

* Hearing loss:
* bilateral symmetrical sensorineural hearing loss
* pure tone thresholds of ≥25 dB HL at one or more frequencies between 250 Hz and 8,000 Hz and differences in thresholds across the two ears of ≤20 dB at every frequency.
* Tinnitus:
* Persistent chronic tinnitus with duration of more than 3 months
* Tinnitus with a Tinnitus Handicap Inventory Grade 2 to 4 (18-76 points)

Exclusion Criteria:

* Non-symmetrical hearing loss
* Raised bi- or multilingually (second language acquired earlier than 6 years of age)
* Women who are currently pregnant or breastfeeding
* History of brain injury or any neurological disorder (y/n)

  • For example, stroke, traumatic brain injury, brain surgery, epilepsy etc.
* Dyslexia
* History of psychiatric disorder
* Recent recreational drug consumption
* Known or suspected drug or alcohol abuse
* Medication with cognitive side effects (e.g., psychoactive medications or sleeping pills)
* Metallic implants in the head region (excluding fixed braces and tooth fillings)
* Any implanted medical device (e.g., cardiac pacemakers)
* Previous enrolment in one of the experiments comprising the main investigational plan

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Experiment 1 - EEG | One study session of 4 hours and 40 minutes
  The primary endpoint is the comparison of neural alpha power lateralization in response to target selection and distractor suppression in individuals with HL, TI and a NH control group.
Experiment 2 - EEG | One study session of 4 hours and 40 minutes
  The primary endpoint is the comparison of the neural tracking of the amplitude envelope of speech between individuals with HL, TI and NH.
Experiment 3 - AAT | One study session of 4 hours and 40 minutes
  The primary endpoint is the comparison of auditory attention performance between tACS over the left temporo-parietal cortex, and an ineffective sham stimulation during and after stimulation relative to pre-stimulation baseline.
Experiment 4 - SAT | One study session of 4 hours and 40 minutes
  The primary endpoint is the comparison of speech comprehension performance between tACS over the left temporo-parietal cortex, and an ineffective sham stimulation during and after stimulation relative to pre-stimulation baseline.
Experiment 5 - EEG 1 | two sessions of 4 hours and 40 minutes on separate days
  The primary endpoint is the comparison of participants' ability to control alpha power lateralization index during training between training conditions (left NF training vs. right NF training).

SECONDARY OUTCOMES:
Experiment 1 - AAT | One study session of 4 hours and 40 minutes
  To test whether alpha power lateralization during distractor suppression and target selection predicts AAT task performance in HL, TI, and NH individuals.
Experiment 2 - SAT | One study session of 4 hours and 40 minutes
  The relation between neural speech tracking and speech comprehension performance in NH, HL, and TI
Experiment 3 - EEG 1 | One study session of 4 hours and 40 minutes
  Comparison of neural alpha power lateralization between stimulation conditions (tACS vs. sham)
Experiment 3 - EEG 2 | One study session of 4 hours and 40 minutes
  Comparison of event-related responses to target and distractor stimuli between stimulation conditions (tACS vs. sham)
Experiment 4 - EEG 1 | One study session of 4 hours and 40 minutes
  Comparison of lateralization index between stimulation conditions (tACS vs. sham)
Experiment 4 - EEG 2 | One study session of 4 hours and 40 minutes
  Comparison between neural tracking of target and distracting speech between stimulation conditions (tACS vs. sham)
Experiment 5 - EEG 2 | two sessions of 4 hours and 40 minutes on separate days
  Comparison of auditory evoked responses to probes presented ipsilateral vs. contralateral to the trained hemisphere
Experiment 5 - EEG 3 | two sessions of 4 hours and 40 minutes on separate days
  Comparison of changes in target and distractor related alpha power lateralization between NF training conditions (left NF training vs. right NF training) pre- vs post NF Training
Experiment 5 - AAT | two sessions of 4 hours and 40 minutes on separate days
  Comparison of auditory attention performance across training conditions (left NF training vs. right NF training)

CONTACTS AND LOCATIONS:
Overall Officials: Basil Preisig, Dr., Principal Investigator — University of Zurich
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The investigators intend to share the raw data of the included participants and the analysis code.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: after the project is completed
Access Criteria: upon personal request